CLINICAL TRIAL: NCT07332455
Title: A Phase 1/2 First-Time-in-Human, Open-label, Multicenter, Dose Escalation and Dose Optimization Study of GSK5471713 in Adult Participants With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: First-Time-in-Human Study of GSK5471713 in Adults With mCRPC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 300164; 2025-523874-17 (Other: EU CT Number)
Record Dates: First submitted 2026-01-09; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms, Prostate
Keywords: Metastatic castration-resistant prostate cancer; First-Time-in-Human; GSK5471713; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants receiving GSK5471713 (Experimental): Participants will receive GSK5471713, according to their allocated dose level guided by the dose escalation study design.
  Interventions: Drug: GSK5471713

INTERVENTIONS:
Drug: GSK5471713 — GSK5471713 will be administered at different dose levels based on the dose escalation study design

SUMMARY:
This first-time-in-human study will evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, preliminary clinical activity, and establish the benefit/risk of GSK5471713 given as a monotherapy in mCRPC.

ELIGIBILITY:
Inclusion Criteria:

* Participants with mCRPC that have histologically or cytologically confirmed adenocarcinoma of the prostate.
* Participants with mCRPC that has prostate cancer progression while on Androgen deprivation therapy (ADT).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
* Progression on ADT and >=1 prior Androgen receptor pathway inhibitors (ARPI) for Hormone-Sensitive Prostate Cancer (HSPC) or Castration resistant prostate cancer (CRPC) and received 1-2 prior taxane based chemotherapy regimens.

Exclusion Criteria:

* Pathological finding consistent with small cell, neuroendocrine carcinoma of the prostate, or any histology different from adenocarcinoma.
* Impaired cardiac function or clinically significant cardiac disease.
* Any significant medical condition, such as uncontrolled infection or clinically significant laboratory abnormality.
* Prior therapy with Androgen receptor (AR) Degrader targeted therapy. Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2028-04-12 (Estimated); Study Completion 2030-04-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) | 28 days
Number of participants with adverse events (AEs), and serious adverse events (SAEs) | Approximately 45 months
Number of participants with adverse events (AEs), and serious adverse events (SAEs) by Severity | Approximately 45 months
Number of participants with AEs leading to dose modifications | Approximately 45 months

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of GSK5471713 | Approximately 45 months
Area under the plasma concentration-time curve from 0 to t (AUC[0-t]) of GSK5471713 | Approximately 45 months
Time to maximum plasma concentration (Tmax) of GSK5471713 | Approximately 45 months
Prostate-specific Antigen Decrease from Baseline >=50% (PSA50) Response Rate | Approximately 45 months
  PSA50 response is defined as a greater than or equal to (>=)50 percent (%) decline in PSA from Baseline, confirmed at least 3 weeks later.
Objective response rate (ORR) per Prostate Cancer Working Group 3 (PCWG3) by investigator assessment | Approximately 45 months
  ORR is defined as the percentage of participants in the ORR Evaluable set who have the Best overall response (BOR) of confirmed Complete response (CR) or Partial response (PR) per PCWG3 guidelines as assessed by investigator.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf